CLINICAL TRIAL: NCT07082127
Title: The Role of Endosymbionts in Trichomonas Vaginalis Pathogenicity
Brief Title: Endosymbionts in Trichomonas Vaginalis Pathogenicity
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Iwona Lesiak-Markowicz, PhD, Medical University of Vienna
Other Study IDs: FWF-ID KLP6210324
Record Dates: First submitted 2025-06-25; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Trichomonas Infection
MeSH Terms: conditions — Trichomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — vaginal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With this project, the investigators aim to expand knowledge on the molecular epidemiology of Trichomonas vaginalis, thereby also evaluating the endosymbionts (Mycoplasma hominis and Trichomonas vaginalis virus) and their impact on T. vaginalis virulence. A key aspect of the study is the direct comparison between identical T. vaginalis isolates harbouring endosymbionts and those from which the endosymbionts have been removed or inhibited. For this purpose T. vaginalis clinical isolates collected in Outpatients' Centre for Infectious Venereal and Dermatological Diseases, Vienna from patients specimens (vaginal swabs or urine) will be tested. Mycoplasma hominis isolates already collected from patients samples will also be analyzed and compared with M. hominis, which are T. vaginalis endosymbionts.

In addition, 700 samples from female sex workers in Austria, who undergo regular medical check-ups, will be examined. The prevalence of sexually transmitted diseases (STDs) will be evaluated using DNA extracted from vaginal swabs, with a particular focus on parasite Trichomonas vaginalis and bacterium M. hominis. Of particular interest is the study of the prevalence of these organisms in a cohort of women who are at increased risk of infection with these pathogens due to their occupation. Moreover, the study will provide detailed information on possible co-infections, as data from routine screenings are available.

DETAILED DESCRIPTION:
For this specific project, patient samples will be cultured in Outpatients' Centre for Infectious Venereal and Dermatological Diseases, Vienna on modified Columbia agar. Specimens will be collected either with a swab, which is then smeared onto the agar plates, or as urine samples, which will be directly spread onto the agar plates. Agar plates that show growth of T. vaginalis after one week of anaerobic incubation at 37°C or M. hominis after two days of anaerobic incubation at 37°C will be set aside. Positive cultures on these agar plates will be collected and transferred to Institute for Specific Prophylaxis and Tropical Medicine (ISPTM) Medical University of Vienna. T. vaginalis and M. hominis isolates will be used for the further characterization. It is planned to remove endosymbionts from the collected T. vaginalis isolates and then test their viability, cytotoxicity, release of pro-inflammatory cytokines and nitric oxide production. M. hominis will be released from T. vaginalis using plasmocin, whereas 2'-C-methylcytidine will be used for Trichomonas vaginalis virus inhibitory assay. The lactase dehydrogenase assay (LDH) will be used to determine cytotoxicity of primary vaginal cells after contact with different T. vaginalis isolates. THP-1 cells (cells derived from leukemia monocytes) will be stimulated with different T. vaginalis isolates and proinflammatory cytokine and nitric oxide production will be evaluated. The expression profiles of putative virulence genes in M. hominis endosymbionts will be also tested. Detection of Ureaplasma spp. DNA in the DNA isolated from T. vaginalis isolates will be performed by PCR and presence confirmed by immunofluorescence and Ureaplasma-specific antibodies.

Vaginal swabs from individual sex-workers (delivered from Austrian Agency for Health and Food Safety) will be used for DNA isolation. For the detection of pathogens, we will use protocols that we have established in our previous studies. Amplified products will be sent for sequencing and compared with reference sequences from GenBank.

ELIGIBILITY:
Inclusion Criteria:

* Trichomonas vaginalis positive samples (vaginal swabs/urine) from Outpatients' Centre for Infectious Venereal and Dermatological Diseases
* female sex-workers subjected to routine testing at Austrian Agency for Health and Food Safety

Exclusion Criteria:

* samples negative for Trichomonas vaginalis from Outpatients' Centre for Infectious Venereal and Dermatological Diseases

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients' Centre for Infectious Venereal and Dermatological Diseases: T. vaginalis positive samples (routine control) Austrian Agency for Health and Food Safety: sex-workers
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Characterisation of T. vaginalis isolates and evaluation of the proportion of sexually transmitted agents in vaginal swabs of Austrian sex workers | 2 years
  Clinical isolates of T. vaginalis or vaginal swabs taken from sex workers will be used in the study.
  Researchers will not have access to any patient information. The results of the experiments conducted on samples from sex workers will be evaluated by sequencing the products obtained by PCR (with primers detecting different sexually transmitted pathogens) and comparing them with the Gene Bank data. In addition, the researchers will assess the percentage of samples positive for T. vaginalis, M. hominis, Ureaplasma spp. among a random group of samples obtained from anonymous sex workers.
  Clinical isolates of T. vaginalis will be tested by PCR for the presence of endosymbionts (M. hominis, T. vaginalis virus). PCR products will also be sequenced and results will be compared with those present in the Gene Bank.

IPD SHARING:
Plan to Share IPD: No